CLINICAL TRIAL: NCT05534789
Title: Clinical Outcomes and Therapy Management Among Patients With Advanced Renal Cell Carcinoma (aRCC) Receiving Systemic First-line (1L) Anti-cancer Treatment Under Daily Routine in Germany: Retrospective Chart Review (RENALISTIC Study)
Brief Title: Treatment Patterns and Clinical Outcomes Among Patients With Advanced Renal Cell Carcinoma (aRCC) Receiving Systemic First-line (1st Line) Anti-cancer Treatment Under Daily Routine in Germany: Retrospective Medical Chart Review (RENALISTIC Study).
Status: Terminated | Type: Observational
Why Stopped: The trial prematurely terminated due to the inability to recruit the planned number of participants. The decision to terminate the trial was not based on any safety and/or efficacy concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A4061099
Record Dates: First submitted 2022-09-06; First posted 2022-09-10 (Actual); Results first posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-11

CONDITIONS: Carcinoma, Renal Cell
Keywords: Real World Chart Review; Retrospective; Germany
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to learn about the treatments used in for advanced renal cell carcinoma as well as effectiveness of these treatments in the real world. Study participants must be:

At least 18 years of age or older. Confirmed renal cell carcinoma Received first line treatment

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with locally advanced or metastatic renal cell carcinoma
* Participants with full medical information is available regarding all treatments before, during and after 1st line

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who received first line treatment for advanced renal call carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A4061099

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of participants with advanced renal cell carcinoma (aRCC) who were greater than or equal to 18 years of age and received first-line (1L) treatment under routine clinical practice in Germany was collected retrospectively from their medical records. Available retrospective data was evaluated/curated per objectives of this study between 15-Oct-2022 to 13-Dec-2023 (approximately 14 months) in the current retrospective observational study.
Groups:
- All Participants: Eligible participants with aRCC who were treated with 1L systemic anticancer treatment in the real world setting under routine clinical practice [started or completed between 01-Jan-2020 to 31-Dec-2021] were included. Data was collected retrospectively for included participants.
Period: Overall Study
Arm/Group | All Participants
Started | 104
Completed | 104
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants who were included in the study.
Groups:
- All Participants: Eligible participants with aRCC who were treated with 1L systemic anticancer treatment in the real world setting under routine clinical practice [started or completed between 01-Jan-2020 to 31-Dec-2021] were included.
Arm/Group | All Participants
Number analyzed (Participants) | 104
Age, Customized [Count of Participants; unit: Participants]
  30-39 years | 1
  40-49 years | 11
  50-59 years | 20
  60-69 years | 40
  70-79 years | 21
  80-89 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 76
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as time from treatment initiation of systemic 1-L therapy start date to documented date of tumor progression or date of death. Disease progression (PD) was defined as greater than equal to (>=) 20% increase in sum of diameters of the target lesions taking as reference the smallest sum on study (this included the baseline sum if that was the smallest on study) or unequivocal progression in non-target lesions or appearance of 1 or more new lesions. Analysis was performed by Kaplan-Meier method.
Time Frame: From treatment initiation date until PD, death or end of follow-up period whichever was earlier (maximum follow-up of 47.1 months)
Population: Analysis population included all eligible participants whose data was retrieved and observed retrospectively in this study.
Measure: Median (Full Range); unit: Months
Arm/Group | All Participants
Number analyzed (Participants) | 104
Months | 9.4 [0.7 to 46.7]

2. Primary Outcome: PFS Rate at Month 6
Description: PFS was defined as time from treatment initiation of systemic 1-L therapy start date to documented date of tumor progression or date of death. Disease progression (PD) was defined as greater than equal to (>=) 20% increase in sum of diameters of the target lesions taking as reference the smallest sum on study (this included the baseline sum if that was the smallest on study) or unequivocal progression in non-target lesions or appearance of 1 or more new lesions. PFS rate was percentage of participants with PFS.
Time Frame: 6 months post treatment initiation date (during maximum follow-up of 47.1 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 104
Percentage of participants | 64.4

3. Primary Outcome: PFS Rate at Month 9
Description: as for outcome 2
Time Frame: 9 months post treatment initiation date (during maximum follow-up of 47.1 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 104
Percentage of participants | 52.9

4. Primary Outcome: PFS Rate at Month 12
Description: as for outcome 2
Time Frame: 12 months post treatment initiation date (during maximum follow-up of 47.1 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 104
Percentage of participants | 41.3

5. Primary Outcome: PFS Rate at Month 18
Description: as for outcome 2
Time Frame: 18 months post treatment initiation date (during maximum follow-up of 47.1 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 104
Percentage of participants | 29.8

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as time from treatment initiation of systemic 1-L therapy to date of death due to any cause or last day of contact. Analysis was performed by Kaplan-Meier method.
Time Frame: From treatment initiation to death due to any cause or last day of contact, whichever occurred first (maximum follow-up of 47.1 months)
Population: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | All Participants
Number analyzed (Participants) | 104
Months | 17.5 [0.3 to 47.1]

7. Secondary Outcome: OS Rate at Months 12 and 18
Description: OS was defined as time from treatment initiation of systemic 1-L therapy to date of death due to any cause or last day of contact. OS rate was measured as percentage of participants alive at specified time points.
Time Frame: 12- and 18-months post treatment initiation date (during maximum follow-up of 47.1 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 104
Percentage of participants
  Month 12 | 65.4
  Month 18 | 49.0

8. Secondary Outcome: Number of Participants According to Different Treatments Received
Description: Number of participants were classified according to different drug groups prescribed: Immune checkpoint inhibitors + Tyrosine kinase inhibitor (ICI +TKI), ICI+ICI, TKI alone and ICI alone.
Time Frame: From treatment initiation to end of follow-up (maximum follow-up of 47.1 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 104
Participants
  ICI + TKI | 48
  ICI + ICI | 21
  TKI alone | 24
  ICI alone | 11

9. Secondary Outcome: Number of Participants With Different Drug Therapies
Description: Number of participants were classified according to different drug regimen therapies prescribed: pembrolizumab + axitinib, nivolumab + ipilimumab, sunitinib, nivolumab, cabozantinib, tivozanib, pembrolizumab, pazopanib, axitinib and avelumab + axitinib.
Time Frame: From treatment initiation to end of follow-up (maximum follow-up of 47.1 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 104
Participants
  Pembrolizumab + Axitinib | 46
  Nivolumab + Ipilimumab | 21
  Sunitinib | 11
  Nivolumab | 8
  Cabozantinib | 6
  Tivozanib | 3
  Pembrolizumab | 3
  Pazopanib | 3
  Axitinib | 1
  Avelumab + Axitinib | 2

10. Secondary Outcome: Best Overall Response
Description: Best overall response was documented as the best response documented in the participant record. CR was defined as complete resolution of all visible disease as per the treating physician's opinion. PR was defined as partial reduction in size of visible disease in some or all areas without any areas of increase in visible disease. Disease progression (PD) was defined as greater than equal to (>=) 20% increase in sum of diameters of the target lesions taking as reference the smallest sum on study (this included the baseline sum if that was the smallest on study) or unequivocal progression in non-target lesions or appearance of 1 or more new lesions. Stable disease was defined as not qualifying for CR, PR, PD. In this outcome measure percentage of participants with best responses are recorded.
Time Frame: From treatment initiation until first documented PD or death or end of follow-up, whichever occurred first (maximum follow-up of 47.1 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 104
Percentage of participants
  CR | 5.8
  PR | 35.6
  SD | 5.8
  PD | 1.9
  Not Evaluable | 5.8
  Not Applicable | 45.2

11. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as time from first disease response (CR/PR) to tumor progression among participants with a documented response and also had a documented date of response. CR was defined as complete resolution of all visible disease as per the treating physician's opinion. PR was defined as partial reduction in size of visible disease in some or all areas without any areas of increase in visible disease. Analysis was performed by Kaplan-Meier method.
Time Frame: From first disease response until tumor progression (maximum follow-up of 47.1 months)
Population: Analysis population included all eligible participants whose data was retrieved and observed retrospectively in this study. Here "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Months
Arm/Group | All Participants
Number analyzed (Participants) | 11
Months | 9.3 [2.1 to 19.8]

12. Secondary Outcome: Time to Progression (TTP)
Description: TTP was defined as time from start of treatment of systemic 1 L therapy up to tumor progression without including deaths. Disease progression (PD) was defined as greater than equal to (>=) 20% increase in sum of diameters of the target lesions taking as reference the smallest sum on study (this included the baseline sum if that was the smallest on study) or unequivocal progression in non-target lesions or appearance of 1 or more new lesions. Analysis was performed by Kaplan-Meier method.
Time Frame: From treatment initiation until tumor progression or end of follow-up whichever occurred first (maximum follow-up of 47.1 months)
Population: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | All Participants
Number analyzed (Participants) | 104
Months | 9.7 [0.7 to 46.7]

13. Secondary Outcome: Time to Next Therapy (TTNT)
Description: TTNT was defined as time from last systemic 1 L therapy administered up to start of next therapy among those participants who completed 1L therapy. Analysis was performed by Kaplan-Meier method.
Time Frame: From last systemic 1 L therapy to start of new therapy (maximum follow-up of 47.1 months)
Population: as for outcome 11
Measure: Median (Full Range); unit: Months
Arm/Group | All Participants
Number analyzed (Participants) | 44
Months | 8.3 [1.4 to 29.9]

14. Secondary Outcome: Number of Participants With at Least 1 Dose Modification or Drug Discontinuation
Description: A dose modification was defined as dose reduction of 1 or all drugs. Number of participants with dose modifications or with an interim/permanent discontinuation of one or all drugs of a therapy were reported in this outcome measure.
Time Frame: From treatment initiation to end of follow-up (maximum follow-up of 47.1 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 104
Participants | 32

15. Secondary Outcome: Number of Participants Continuing Therapy After Dose Modification
Description: A dose modification was defined as dose reduction of 1 or all drugs. Number of participants with dose modification of one or two drugs but continuing therapy were reported in this outcome measure.
Time Frame: From treatment initiation to end of follow-up (maximum follow-up of 47.1 months)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 32
Participants | 23

16. Secondary Outcome: Number of Participants With Discontinuation of One or Two Drugs
Description: Number of participants with discontinuation of one or two drugs were reported in this outcome measure.
Time Frame: From treatment initiation to end of follow-up (maximum follow-up of 47.1 months)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 32
Participants | 9

17. Secondary Outcome: Number of Participants Continuing Therapy After Temporary/Permanent Discontinuation of Single Drugs
Description: Number of participants continuing therapy after temporary/permanent discontinuation of single drugs are reported in this outcome measure.
Time Frame: From treatment initiation to end of follow-up (maximum follow-up of 47.1 months)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 9
Participants | 1

ADVERSE EVENTS:
Time Frame: All-cause mortality: From treatment initiation to end of follow-up (maximum follow-up of 47.1 months). Data for non-serious adverse events (non-SAE) and serious adverse events (SAEs) were not collected and evaluated during the study; hence timeframe is not applicable for non-SAEs and SAEs
Description: This study is retrospective, it involves data that exist as structured data by the time of study start. From data source, individual participant data were not retrieved or validated. The minimum criteria for reporting an adverse event (AE) (identifiable participant, identifiable reporter, a suspect product, and event) cannot be met. The customized CRF did not collect data on adverse events. There was no collection of adverse events in the study, hence results for them are not recorded.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 36/104
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT05534789/Prot_SAP_000.pdf